CLINICAL TRIAL: NCT02016313
Title: Evaluation of the Effect of Cervical Spine Treatment in Tinnitus Patients
Brief Title: The Effect of Physiotherapy on Cervicogenic Somatic Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Sarah Michiels, Assistent Rehabilitation Sciences and Physical Therapy, Universiteit Antwerpen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: G850-tinnitus1
Record Dates: First submitted 2013-12-09; First posted 2013-12-19 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate therapy (Experimental): Physiotherapy protocol
  Interventions: Other: physiotherapy
- waiting list (Placebo Comparator): Physiotherapy protocol
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: physiotherapy

SUMMARY:
The purpose of this study is to determine whether physiotherapy is effective in the treatment of a group of tinnitus patients with neck complaints.

ELIGIBILITY:
Inclusion Criteria:

* severe chronic non-fluctuating subjective cervicogenic somatic tinnitus, which has been stable for at least three months, combined with neck complaints

Exclusion Criteria:

* objective tinnitus
* subjective tinnitus with etiologies, such as hearing loss or Meniere's disease, severe depression (> 19 on the Beck depression questionnaire)
* progressive middle ear pathology
* intracranial pathology
* traumatic cervical spine injury
* tumors
* cervical spine surgery
* any cervical spine condition in which physical therapy treatment is contra- indicated
* received physical therapy treatment directed to the cervical spine in the past 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Tinnitus Functional Index | pre treatment, post treatment, 6 and 12 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Paul Van de Heyning, PhD, MD, Study Chair — Universiteit Antwerpen; Willem De Hertogh, PhD, Study Chair — Universiteit Antwerpen
Locations (1):
- University Hospital of Antwerp, Edegem, Antwerp, Belgium

REFERENCES:
- [Derived] Michiels S, Van de Heyning P, Truijen S, Hallemans A, De Hertogh W. Does multi-modal cervical physical therapy improve tinnitus in patients with cervicogenic somatic tinnitus? Man Ther. 2016 Dec;26:125-131. doi: 10.1016/j.math.2016.08.005. Epub 2016 Aug 26. PMID 27592038
- [Derived] Michiels S, De Hertogh W, Truijen S, Van de Heyning P. Physical therapy treatment in patients suffering from cervicogenic somatic tinnitus: study protocol for a randomized controlled trial. Trials. 2014 Jul 22;15:297. doi: 10.1186/1745-6215-15-297. PMID 25056151